CLINICAL TRIAL: NCT06506825
Title: The Fourth Hospital of Hebei Medical University
Brief Title: Construction and Application of Database of Hebei Provincial Gastric Cancer Collaborative Network Driven by Artificial Intelligence Technology
Status: Recruiting | Type: Observational
Sponsor: Qun Zhao (Other)
Responsible Party: Sponsor-Investigator, Qun Zhao, Professor, Hebei Medical University
Organization: Hebei Medical University (Other)
Other Study IDs: HBGCCN
Record Dates: First submitted 2024-07-12; First posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: The Study Focuses on Gastric Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Gastric Cancer AI-driven Data Integration Genomic Analysis Biomarker — Enter the clinical and related test, examination and treatment information of all gastric cancer patients, and find risk factors that affect the prognosis

SUMMARY:
This clinical trial aims to construct and apply a collaborative network database for gastric cancer in Hebei Province, driven by artificial intelligence (AI) technology. The project seeks to integrate clinical data, genomic information, and treatment outcomes from multiple hospitals and research centers within the region. By leveraging advanced AI algorithms, the database will facilitate comprehensive data analysis to identify novel biomarkers, optimize therapeutic strategies, and improve patient outcomes. This initiative will also support real-time data sharing and collaboration among healthcare providers, researchers, and policymakers, ultimately enhancing the overall management and treatment of gastric cancer in Hebei Province.

ELIGIBILITY:
Inclusion Criteria:

All patients with gastric cancer

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients with gastric cancer
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
5-year overall survival | 2025-12-31
  5-year overall survival

SECONDARY OUTCOMES:
5-year recurrence-free survival | 2025-12-31
  5-year recurrence-free survival

CONTACTS AND LOCATIONS:
Locations (1):
- Department of General Surgery, Shijiazhuang, Hebei, China